CLINICAL TRIAL: NCT03380299
Title: Association of CD49d and CD44 in CLL Patients and Their Role in Prognosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ALShymaa faheem solyman ali, RESIDENT DOCTOR, Assiut University
Other Study IDs: 1700258
Record Dates: First submitted 2017-12-08; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Cellular Diagnosis, Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The interactions of chronic lymphocytic leukemia cells with the microenvironment in secondary lymphoid tissues and the bone marrow are known to promote CLL cell survival and proliferation

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most common type of chronic leukemia, accounting for approximately 40% of all leukemia's and mainly affecting older individuals. As it has a highly variable clinical course, identification of molecular and biological prognostic markers has provided new insights into the risk stratiﬁcation of patients with CLL .

The interactions of chronic lymphocytic leukemia cells with the microenvironment in secondary lymphoid tissues and the bone marrow are known to promote CLL cell survival and proliferation . CD49d (one of biomarkers) is one of independent prognostic risk parameter in CLL with important roles in shaping these interactions.

CD49d also is one of independent prognostic risk parameters in CLL that predict adverse outcome and linked to processes involved in interaction with the vascular endothelium and/or migration into the extravascular compartments .

The cell-surface glycoprotein CD44 is involved in cell motility, cellular trafficking, and stem cell differentiation . It contributes to the phenotypic hallmarks of many cancers, such as invasiveness, self-renewal, and sustained survival. CD44 transmits both growth and apoptotic signals, a functional duality that is also observed in hematologic malignancies.

CD44 expression in CLL is mediated by the tumor microenvironment. As a coreceptor, CD44 promotes leukemogenesis by regulating stimuli of MCL1 expression. Moreover, CD44 can be addressed therapeutically in CLL by specific antibodies.

ELIGIBILITY:
Inclusion Criteria:

* All patients are newly diagnosed as CLL

Exclusion Criteria:

* : patients with associated malignancies

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 30 patients All patients are newly diagnosed as CLL patients with associated malignancies
  * Clinical history and clinical examination by the physician.
  * Complete blood picture: on peripheral blood sample.
  * BM aspiration: allowing diagnosis of the type of leukemia.
  * Immunophenotyping by flowcytometer: will be done on peripheral blood or bone marrow aspirate specimens for establishing diagnosis of CLL by detecting its markers ( CD5,CD19,CD23) and for detecting membrane expression of CD49d and CD 44
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2016-07-14 (Actual); Primary Completion 2018-09-14 (Estimated); Study Completion 2018-12-14 (Estimated)

PRIMARY OUTCOMES:
To what extent the identiﬁcation of molecular and biological prognostic markers has provided new insights into the risk stratiﬁcation of patients with CLL . | 1 YEAR
  detecting membrane expression of CD49d and CD 44 and thier role in prognosis of CLL patients.